CLINICAL TRIAL: NCT01212003
Title: Natural History of Tuberculosis
Brief Title: Training Protocol on the Natural History of Tuberculosis
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100195; 10-I-0195
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-27

CONDITIONS: Mycobacterium Infections; Tuberculosis, Multidrug-Resistant; Latent Tuberculosis; Tuberculosis; Extensively Drug-Resistant Tuberculosis
Keywords: TB; Mycobacterium Tuberculosis; Active Tuberculosis; Latent Tuberculosis; MDR TB; Natural History; Tuberculosis
MeSH Terms: conditions — Mycobacterium Infections; Tuberculosis, Multidrug-Resistant; Latent Tuberculosis; Tuberculosis; Extensively Drug-Resistant Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active TB: subjects with active TB as determined by smear, culture, or biopsy or have appropriately documented clinically suspicious active TB without definitive microbiology confirmation
- Latent TB: subjects with documented evidence of a positive PPD skin test or Interferon Gamma Release Assays (IGRA) test meeting American Thoracic Society (ATS)/CDC guidelines for latent TB

SUMMARY:
Background:

- Tuberculosis (TB) is an infectious disease that affects numerous people worldwide. Researchers are interested in actively recruiting individuals with TB for research and treatment studies.

Objectives:

- To collect blood and other samples to study the natural history of tuberculosis.

Eligibility:

- Individuals 2 years of age and older who have either active or latent tuberculosis.

Design:

* Latent TB patients: Participants will have a single study visit with a physical examination and medical history, and will provide blood samples for testing.
* Active TB patients: Participants will have an initial visit with a physical examination and medical history, and will provide blood samples for testing. Participants will also provide sputum samples if required, and may have an optional skin punch biopsy to collect a sample of skin tissue for study.
* Treatment for active TB will be provided as part of this protocol.
* Active TB participants may be asked to return for study visits every 1-2 months while receiving treatment....

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (MTB) is a slow-growing bacterium that establishes latent infection in millions of persons worldwide, but only leads to disease in 10% or less of these individuals. It typically causes pneumonia, however dissemination to almost any other organ is possible. Drug resistance of the organism, co-infection with HIV, and paradoxical reactions upon treatment are all factors that may complicate treatment.

Host defense against mycobacterial infections is important. Specific defects within the innate immune system lead to Mendelian susceptibility to mycobacterial infections. HIV infected individuals and persons treated with anti-tumor necrosis factor antibodies are highly susceptible to tuberculosis (TB) infection. Genetic influence on susceptibility to TB disease is complex and does not seem to be confined to a single gene or pathway.

Advancement in molecular techniques has expanded our understanding of the pathogenesis and epidemiology of MTB. Identification of gene mutations that confer antibiotic resistance are being exploited as alternatives to conventional drug susceptibility testing.

The natural history of all forms of TB disease (including co-infection with HIV and other infections) will be followed, and MTB isolates and blood from 100 infected patients will be obtained in order to study organism virulence and host immune function and genetic/epigenetic factors. While it is recognized that the number of TB cases that occur in the Washington, DC area and nationally is low, it is imperative that a mechanism is in place to evaluate and treat these patients at the NIH Clinical Center. This protocol will also allow NIH infectious diseases trainees to manage challenging cases of TB.

ELIGIBILITY:
* INCLUSION CRITERIA:

FOR ALL PATIENTS

Patients may be included in this study who:

* Have or are suspected to have TB infection.
* Are aged 2 years or older.
* Have a primary care physician, infectious diseases physician, pulmonologist, or TB specialist outside of the NIH who can provide care of his or her TB infection outside the NIH, provide directly observed therapy (DOT) if necessary, and monitor for side effects and toxicity of TB medications.
* Are willing to consent to storage of specimens for future research.
* Able to provide informed consent for themselves or, if they lack the capacity to provide informed consent, have an appropriate Legally Authorized Representative (LAR; the study team will comply with NIH Human Research Protection Program [HRPP] Policy 403).

FOR PATIENTS WITH LATENT TB

In addition to the above-described inclusion criteria for all patients, patients may be included in the Latent TB part of this protocol who:

-Have documented evidence of a positive purified protein derivative (PPD) skin test or Interferon-gamma Release Assays (IGRA) test meeting American Thoracic Society (ATS)/CDC guidelines for latent TB; conversion can have occurred at any time.

FOR PATIENTS WITH ACTIVE TB

In addition to the above-described inclusion criteria for all patients, patients may be included in the Active TB part of this protocol who:

* Have active TB of any drug susceptibility pattern and any site of infection as determined by smear, culture, or biopsy.
* Have appropriately documented clinically suspicious active TB without definitive microbiology confirmation.

EXCLUSION CRITERIA:

Patients will be excluded from this study who:

* Are incarcerated.
* Have been ordered by a court to take TB medications.
* Are unwilling or unable to comply with prescribed therapy.
* Are pregnant.

EXCLUSION OF SPECIFIC POPULATIONS

Children: Children under the age of 2 are not eligible to enroll. The addition of the very young will not provide enough additional insights to justify the risk to this specific population.

Pregnant women: Pregnant women are not eligible for participation in this protocol because the study objectives can be achieved without the enrollment of this population. Enrolled participants who become pregnant during the study will be withdrawn.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be referred by their physicians for study participation. In many cases, participants will be referred by physicians at their local health department tuberculosis clinics (where they often receive DOT for TB treatment). Family members may be recruited through requests made by the index case that family members contact study personnel for participation. A patient can be referred at any time point while he or she is receiving active treatment for tuberculosis. Male and female patients will be accepted without preference. Patients age 2 and older are eligible; however, severe infections may require highly specialized pediatric teams and institutions. Some referrals of pediatric cases will not be able to be handled appropriately at the NIH and may be deemed ineligible for admission, as determined by the Principal Investigator (PI). NIH employees and members of their immediate families may participate in this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Increase in the number of TB patients being actively followed at the NIH CC to provide information on TB patients with DS and drug-resistant disease for hypothesis generation and hands-on experience in the management of TB | ongoing
  increased number of TB patients being actively followed at the NIH CC

SECONDARY OUTCOMES:
Determination of subsets of lymphoid populations during various points in the treatment of TB | ongoing
  subsets of lymphoid populations during various points in treatment of TB
Description of whole genome sequences and their possible relationship to TB infection | ongoing
  possible relationship of whole genome sequences to TB infection
Collection of MTB specimens for studies of the organism and its pathogenesis | ongoing
  collection of MTB specimens

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenzweig SD, Holland SM. Defects in the interferon-gamma and interleukin-12 pathways. Immunol Rev. 2005 Feb;203:38-47. doi: 10.1111/j.0105-2896.2005.00227.x. PMID 15661020
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-I-0195.html